CLINICAL TRIAL: NCT00457028
Title: Efficacy of Treatment for Obsessive Compulsive Disorder
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Maureen Whittal, University of British Columbia
Other Study IDs: H03-80266
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Anxiety; Treatment efficacy
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of these questionnaires is to give us an overview of how OCD has affected your life and perhaps also to give us some clues about things that may have set you up to experience OCD.

DETAILED DESCRIPTION:
For us to evaluate the efficacy of our treatment programs, we are interested in your responses before and after treatment. We use two methods to evaluate the efficacy of our treatments: questionnaires and interviews with a member of the Anxiety Disorders Clinic. As part of standard clinic procedure, each person in the program completes an in-person interview with a staff member who will determine your suitability for treatment. If you have received this questionnaire packet, it is likely that your concerns will be appropriately addressed in the Anxiety Disorders Clinic. The purpose of the questionnaire packet is to assess the severity of your obsessive-compulsive disorder; its impact on your functioning, and factors that may contribute to the onset or maintenance of your OCD (e.g., depression, personal standards). We will ask you to complete this questionnaire again when you have completed your treatment along with a brief telephone interview with a staff member of the Anxiety Disorders Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Anxiety Disorders Clinic who receive a primary diagnosis of Obsessive Compulsive Disorder, and are accepted for treatment at the clinic.

Exclusion Criteria:

* Individuals who either have not sought treatment for anxiety at the Anxiety Disorders Clinic or patients who did not receive a primary diagnosis of Obsessive Compulsive Disorder.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the study will be recruited from individuals receiving treatment at the Anxiety Disorders Clinic of UBC Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2003-05; Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Whittal, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Anxiety Disorders Clinic, University of British Columbia, Vancouver, British Columbia, Canada